CLINICAL TRIAL: NCT01320475
Title: Thoracic Epidural Analgesia: Epidural Levobupivacaine and Sufentanil Versus Epidural Levobupivacaine and Intravenous Ketamine
Brief Title: Epidural Levobupivacaine-sufentanil Versus Epidural Levobupivacaine and Intravenous Ketamine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty of Recruitment
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009/04
Record Dates: First submitted 2011-03-19; First posted 2011-03-22 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Thoracic Surgery
Keywords: thoracic epidural analgesia; epidural opioid; ketamine; adverse effect
MeSH Terms: interventions — Sufentanil; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- iv Ketamine (Experimental): Epidural infusion of levobupivacaine and saline (placebo for sufentanil)and iv infusion of ketamine Up to the third postoperative day (6 PM)
  Interventions: Drug: Ketamine
- Sufentanil (Active Comparator): Epidural infusion of levobupivacaine (1,25 mg/ml) and sufentanil(1 ml = 50 µg diluted in the 200 ml bag of levobupivacaine) IV infusion of saline (placebo for ketamine)
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Sufentanil — Epidural infusion of levobupivacaine (1,25 mg/ml) and sufentanil(1 ml = 50 µg diluted in the 200 ml bag of levobupivacaine) IV infusion of saline (placebo for ketamine)
  Arms: Sufentanil
Drug: Ketamine — Epidural infusion of levobupivacaine (1,25 mg/ml) and saline (1 ml = 50 µg diluted in the 200 ml bag of levobupivacaine) IV infusion of ketamine (2 µg/kg/minute) Up to the third postoperative day (6 PM)
  Arms: iv Ketamine

SUMMARY:
Thoracic epidural analgesia is often proposed to thoracotomized patients. A local anesthetic and an opioid are generally associated to produce an epidural analgesia. However, opioid epidural administration is frequently associated with adverse effects as nausea, vomiting, urinary retention, ... On the other hand, iv ketamine has been demonstrated to be an effective analgesic.

The purpose of the study is to compare the epidural administration of levobupivacaine and sufentanil or the epidural administration of levobupivacaine associated with the iv administration of ketamine.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 yrs
* class ASA I, II or III
* lung surgery

Exclusion Criteria:

* Contra-indication to the achievement of epidural analgesia
* Preoperative chronic pain,
* Contra-indication to ketamine
* Hypersensitivity to ketamine or any excipients
* Uncontrolled hypertension,
* Stroke
* Heart failure
* Hepatic porphyria
* Contra-indication to sufentanil
* Hypersensitivity to sufentanil, opioids or any excipients
* Treatment with an opioid agonist-antagonist,
* Contra-indication to levobupivacaine
* Hypersensitivity to levobupivacaine, local anesthetics of the amide or any excipients
* Hypotension, shock

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of an adverse event due to the analgesic protocol | one week
Efficacy of the analgesic regimen | third postoperative day

SECONDARY OUTCOMES:
postoperative rehabilitation | two weeks
postoperative complications (pulmonary, others) | one month
length of stay | one month
patient's satisfaction | sortie de l'hopital
Occurence of a chronic pain | end the first postoperative year

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Foch, Suresnes, France